CLINICAL TRIAL: NCT04091607
Title: An Evaluation of Pain, Anxiety, Desire for Repeat Procedure, and Satisfaction Utilizing Music Therapy for Chronic Low Back Pain Patients During Lumbar Medial Branch Blocks"
Brief Title: Using Music During Lumbar Medial Branch Block Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00060053
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Lower Back Pain; Lumbar Spondylosis
Keywords: lumbar medial branch block; chronic back pain; lower back pain; lumbar spondylosis
MeSH Terms: conditions — Low Back Pain; Spondylosis | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Group 1 will listen to Music during the procedure. Group 2 will not hear any music during the procedure
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy Intervention Group (Active Comparator): listen to preferred choice of music during the Lumbar Medial Branch Block procedure.
  Interventions: Other: Music Therapy
- Control Group (No Intervention): No music will be provided but will be provided earbuds. The sound environment will be standard for procedures by closing procedure room door and minimizing extraneous sounds.

INTERVENTIONS:
Other: Music Therapy — Subject will listen to Music using provided ear buds or headphones.
  Arms: Music Therapy Intervention Group

SUMMARY:
The purpose of this study is to determine if music therapy during interventional lumbar medial branch blocks for chronic lower back pain will lower pain scores and anxiety levels, while increasing patient desire for repeat procedure as well as patient satisfaction.

DETAILED DESCRIPTION:
Subjects will be put into 1 of 2 groups, Music or the Control Group (no music). The music group will listen to patient's preferred music on Pandora station broadcast using Headphones or Wireless Earbuds with Tablet or Computer. Hearing impaired patients will have an option of non-earbud headphones. . Earbuds or headphones will be used regardless of music therapy playing. . The control group will be provided earbuds or alternative headphone as well, however, with no music. The sound environment will be standardized for procedure by closing procedure room door and minimizing extraneous sounds (i.e. from equipment, alarms, etc.,).

ELIGIBILITY:
Inclusion Criteria:

* Age> or equal to 18
* History of documented chronic lower back pain

Exclusion Criteria:

* Patient refusal
* Deafness (unless corrected with a hearing aid)
* Initial Pain Score < 3
* Prior Lumbar Medial Branch Blocks/Radiofrequency ablation therapy
* Any woman who is currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Pain Scores with True Visual Analog scale | Day 1 Pre Procedure
  Score ranges from 0 to 10 with higher score denoting more pain.
Pain Scores with True Visual Analog scale | Day 1 Post Procedure
  Score ranges from 0 to 10 with higher score denoting more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Columbano, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04091607/ICF_000.pdf